CLINICAL TRIAL: NCT04970914
Title: Anlotinib Hydrochloride In Combination With Penpulimab (AK105) in Patients With Chemo-refractory Metastatic Colorectal Cancer, Open, Single Arm,Exploratory Clinical Trial(ALTER-C003)
Brief Title: Anlotinib Plus Penpulimab (AK105) for Chemo-refractory Metastatic Colorectal Cancer:ALTER-C003
Acronym: ALTER-C003
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, YueJuan Cheng, Prof.M.D., Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-2986B
Record Dates: First submitted 2021-07-05; First posted 2021-07-21 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — anlotinib; penpulimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib+Penpulimab (Experimental)
  Interventions: Drug: Anlotinib; Drug: Penpulimab

INTERVENTIONS:
Drug: Anlotinib — 12mg, continuous oral 2 weeks stop for 1 week, 21 days for a treatment cycle.
  Other Names: anlotinib hydrochloride
Drug: Penpulimab — Penpulimab 200 mg administered intravenously every 3 weeks.
  Other Names: AK105

SUMMARY:
A single-arm, open-label clinical trial, focus on the safety and efficacy of anlotinib hydrochloride in combination with Penpulimab (AK105) in patients with Chemo-refractory Metastatic Colorectal Cancer (mCRC)

ELIGIBILITY:
Inclusion Criteria:

* Patients participate in the study voluntarily and sign informed consent with good compliance.
* Be 18 years of age or older on day of signing informed consent.
* Histological or cytological confirmation of Metastatic Colorectal Cancer(T1-4N0-2M1).
* At least one measurable lesion, with diameter ≥ 10mm measured by spiral MRI/CT scan per RECIST1.1.
* Participants must have received and progressed through or become intolerant to fluoropyrimidine, irinotecan, oxaliplatin, Exceptions may apply.
* Eastern Cooperative Oncology Group Performance Status 0 or 1.
* Life expectancy of at least 3 months.
* Main organs function is normal. (normal main organs function as defined below: Hemoglobin (Hb) ≥ 90 g/L, Neutrophils (ANC) ≥ 1.5×109/L, leucocyte (WBC) ≥ 3.0×109/L,Platelet count (PLT) ≥ 75×109/L,Total bilirubin (TBIL) ≤ 1.5 × normal upper limit (ULN), Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 2.5 ×ULN, If liver metastasis is present，ALT and AST<5ULN ；Serum creatinine (Cr) ≤ 1.5× ULN or Creatinine Clearance rate(CCr) ≥60ml/min，Doppler ultrasound evaluation: left ventricular ejection fraction (LVEF) > 50%)
* The woman patients of childbearing age who must agree to take contraceptive methods (e.g. intrauterine device, contraceptive pill or condom) during the research and within another 3 months after it; who are not in the lactation period and examined as negative in blood serum test or urine pregnancy test within 7 days before the research; The man patients who must agree to take contraceptive methods during the research and within another 8 weeks after it.

Exclusion Criteria:

* Histological or cytological confirmation of mucinous adenocarcinoma or ovarian transcoelomic metastasis
* Patients who had previously received treatment with Anlotinib or anti-programmed cell death protein 1 (PD-1), programmed cell death protein 1 ligand 1 (PD-L1), or cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) inhibitors other immunotherapy against .
* Patients who had previously received treatment within 2 weeks or Participated in other anti-tumor clinical trials within 4 weeks.
* Patients with a large amount of pleural effusion or ascites requiring drainage.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
* Patients who underwent major surgery within 4 weeks.
* Regardless of the severity, patients with any physical signs or history of bleeding, patients with bleeding or bleeding events greater than or equal to CTCAE 3 within four weeks prior to the first administration, or patients with unhealed wounds, fractures, ulcers.
* Patients with a risk of gastrointestinal bleeding may not be enrolled.
* Patients with arterial or venous thromboembolic events occurred within 6 months, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis and pulmonary embolism.
* Patients with any severe and/or unable to control diseases，including： Patients with unsatisfactory blood pressure control using antihypertensive drugs (systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥100) mmHg); Patients with Grade 2 or higher myocardial ischemia, myocardial infarction or malignant arrhythmias(including male QTc≥450ms; female QTc≥470ms) and patients with Grade 2 or higher congestive heart failure (NYHA Classification); Patients with active or unable to control serious infections, which is over level 2 in CTC AE (4.0); Patients with poorly controlled diabetes (fasting blood glucose(FBG)>10mmol/L); Patients with kidney failure who require hemodialysis or peritoneal dialysis; Patients with interstitial lung disease with symptoms or signs of activity；Patients with a history of immunodeficiency, including a positive HIV test or other acquired, congenital immunodeficiency disease, or a history of organ transplantation; Urine routine indicates that urine protein ≥ ++, and confirmed 24-hour urine protein quantitation > 1.0 g; Patients with any of the following coagulation functions are abnormal, including: Prothrombin time (PT)>ULN+4s, Activated partial thromboplastin time (APTT) >1.5ULN s, international normalized ratio (INR)>1.5; Patients with a seizure disorder who require pharmacotherapy.
* Patients who have got non remissive toxic reactions derived from any treatment, which is over level 1 in CTC AE (4.0).
* Has a diagnosis of immunodeficiency or is receiving chronic steroid therapy of prednisone ≥ 10 mg daily or any equivalent dose of corticosteroids.
* Has received a live vaccine or attenuated vaccine within 30 days prior to trial registration.
* Symptoms that affect oral medication and cannot be controlled through proper treatment (such as inability to swallow, chronic diarrhoea and intestinal obstruction, etc.).
* Female patients who are pregnant or breastfeeding.
* Patients with drug abuse history and unable to get rid of or patients with mental disorders.
* Patients who had serious adverse effect to Anlotinib or Penpulimab or any of its excipients
* Known hypersensitivity to other Monoclonal Antibody or any of its excipients.
* Patients with concomitant diseases which could seriously endanger their own safety or could affect completion of the study according to investigators' judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-11-05 (Actual); Primary Completion 2022-08-23 (Estimated); Study Completion 2023-08-23 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | up to 24 months
  Progression-free Survival (PFS) (median) was determined using the number of months measured from the initial date of treatment to the date of documented progression, or the date of death (in the absence of progression) of participants. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | up to 24 months
  Objective response rate is defined as the percentage of subjects whose best response was complete response (CR) or partial response (PR) according to the RECIST v1.1
Disease Control Rate (DCR) | up to 24 months
  Disease control rate is defined as the percentage of subjects whose best response was CR, PR or stable disease (SD) according to the RECIST v1.1.
Duration of Response (DOR) | up to 24 months
  Duration of Response is defined as the percentage of subjects whose best response was CR, PR or stable disease (SD) according to the RECIST v1.1 or death due to any cause, whichever occurs first.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Until 30 day safety follow-up visit
  Adverse events assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (version 5.0).
Overall Survival (OS) | Up to 24 months
  Overall Survival (OS) (median) is determined using the number of months measured from the initial date of treatment to the recorded date of death of participants.

OTHER OUTCOMES:
Number of TB cells count and interleukin-6/8/10 | through study completion, an average of 2 year
  Objectives to analyse the subsets of TB cells and interleukin-6/8/10 associated treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jianfeng Zhou, Principal Investigator — Peking Union Medical College Hospital
Locations (8):
- China (8):
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - China-Japan friendship hospital, Beijing, Beijing Municipality
  - Hebei Petro China Central Hospital, Langfang, Hebei
  - The Fourth Hospital of Hebei Medical University (Hebei Cancer Hospital), Shijiazhuang, Hebei
  - General Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - Peking Union Medical College Hospital, Beijing
  - The First Hospital Of China Medical University, Shenyang
  - The People's Hospital Of Liaoning Province, Shenyang

IPD SHARING:
Plan to Share IPD: No